CLINICAL TRIAL: NCT00658749
Title: A Phase 1, Single-Center, Randomized, Double-Blind, Placebo-Controlled Study of AIR645 in Healthy Subjects and Subjects With Controlled Asthma
Brief Title: A Phase 1 Study of AIR645 in Healthy Subjects and Subjects With Controlled Asthma
Acronym: AIR645-CS1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Altair Therapeutics, Inc. (Industry)
Responsible Party: Susan Gregory/Chief Scentific Officer, Altair Therapeutics, Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AIR645-CS1
Record Dates: First submitted 2008-04-11; First posted 2008-04-15 (Estimated); Last update posted 2009-06-25 (Estimated); Status verified 2009-06

CONDITIONS: Asthma
Keywords: AIR645; Altair Therapeutics; IL4; IL13; IL-4; IL-13
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): AIR645 (an IL-4/IL-13 dual cytokine signaling inhibitor) solution (diluent: physiologic saline solution)
  Interventions: Drug: AIR645
- 2 (Placebo Comparator): Physiologic saline solution
  Interventions: Drug: Physiologic saline solution

INTERVENTIONS:
Drug: AIR645 — AIR645 (blinded) by nebulization, range of doses, maximum of one dose per day, maximum of 6 doses in 22 days.
  Arms: 1
Drug: Physiologic saline solution — Placebo (blinded) by nebulization, range of doses, maximum of one dose per day, maximum of 6 doses in 22 days.
  Arms: 2

SUMMARY:
This is a phase one study to evaluate the safety, tolerability, and bioavailability of nebulized AIR645.

ELIGIBILITY:
Inclusion Criteria*:

* Good General Health (with or without allergic rhinitis and/or controlled asthma)
* Non-smoker for at least 2 years
* Normal lung function (DLCO)
* Able to provide informed consent and to understand and comply with the requirements of the study

Exclusion Criteria*:

* Clinically significant medical history or condition which precludes participation
* Clinically significant ECG abnormality
* Clinically significant VS or PE abnormality
* Clinically significant screening lab abnormality
* Abnormal lung function (FEV1 <80% predicted)
* Respiratory infection within 14 days of randomization
* HBV, HCV, or HIV
* Breastfeeding or pregnant female
* History of alcohol abuse or illicit drug use within past 24 months
* Use of any tobacco or nicotine-containing product within past 6 months
* Use of any herbal supplement, over-the-counter drug, or prescription drug that is not allowed per protocol
* Use of any investigational drug within past 30 days
* Use of any investigational monoclonal antibody or recombinant protein within past 90 days
* Donation of plasma within past 7 days
* Donation or loss of whole blood within past 56 days

  * Simplified list of I/E criteria; unabridged list available upon request.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-04; Primary Completion 2009-04 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Measures of the safety and tolerability of AIR645 include documentation of adverse events and changes (compared to baseline) in vital signs, physical examination, pulmonary function tests, heart rhythm, and laboratory tests. | During dosing and for two weeks after dosing

SECONDARY OUTCOMES:
Bioavailability | During dosing and for two weeks after dosing

CONTACTS AND LOCATIONS:
Overall Officials: Mike Hodges, MD, Study Director — Altair Therapeutics
Locations (1):
- Contract Research Organization (CRO) appointed by Altair Therapeutics--Altair's offices are in:, San Diego, California, United States